CLINICAL TRIAL: NCT04915599
Title: Pilot Trial for Feasibility and Patient Reported Tolerance of Cryo-therapy With the Cooral ® Mouth Cooling Device [MCD) in Patients Undergoing Radiation Therapy for Head and Neck Malignancies
Brief Title: Feasibility and Patient Reported Tolerance of Cryotherapy With the Cooral ® Mouth Cooling Device [MCD) in Patients Undergoing Radiation Therapy
Acronym: CooRay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2021-00887; th21Bunea
Record Dates: First submitted 2021-05-26; First posted 2021-06-07 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Oral Mucositis
Keywords: Cooral ® Mouth cooling device (MCD); cryotherapy; radiation therapy; severe oral Mucositis; Head and Neck Cancer; Mouth Cooling Device
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Patients are assigned to using the Cooral® MCD after radiotherapy for 60 min. along with general oral care (GOC). The MCD will be placed into the subjects' mouth and remain intraorally for 60 minutes. After each fraction, i.e. session of RT, the subjects insert the MCD inside their mouth and can start the Cooral ® thermostat system themselves when they feel comfortable. The stopwatch will be started by the patient as soon as thermostat is running. The patient is asked to write down the starting and the stopping time of the 60-minute procedure. Thereafter the subject will receive a questionnaire to record the tolerance for the device. Patients will be also informed about standard of care (SOC) that should be regularly performed.
  Interventions: Device: Cooral® mouth cooling device (MCD)

INTERVENTIONS:
Device: Cooral® mouth cooling device (MCD) — Cooral® mouth cooling device (MCD) to prevent oral mucositis (QM) in patients undergoing radiation therapy for head and neck malignancies

SUMMARY:
This study is to investigate the use of the Cooral ® standardized CyT device to achieve a constant and reproducible cooling of the oral mucosa to prevent OM in patients undergoing RT in the head and neck region.

DETAILED DESCRIPTION:
Severe oral mucositis (SOM) is a major side-effect during (chemo)-radiation of malignancies of the head and neck. There is no standard management of SOM. Previous studies have shown an effect of cryotherapy (CyT) on the incidence and duration of SOM in chemotherapy patients. Especially in palliative cases it is necessary to keep treatment related morbidities low.

Due to the difficulties and possible side effects of ice chips (IC), a closed system, such as an intra oral mouth cooling device (MCD) might help to fully unfold the efficacy of CyT in the prevention of radiation therapy (RT)-induced oral mucositis (OM), without putting the patient at risk for infections.The Cooral ® system, provided by a Swedish medical technology company free of charge, is composed of two parts: 1) the Cooral ® system itself, which is a portable thermostat allowing to adjust temperatures , ranging between 6 and 22°C. 2) the mouthpiece composed of flexible plastic material (polyolefin polymer compound based on ethylene-vinyl acetate copolymer) that is connected via two flexible plastic hoses to the Mouth Cooling Device (MCD). The water cooled inside the thermostat then circulates through the mouthpiece, allowing the mucosa to be cooled continuously and keep the desired temperature for any time.

This study is to investigate the use of the Cooral ® standardized CyT device to achieve a constant and reproducible cooling of the oral mucosa to prevent OM in patients undergoing RT in the head and neck region.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score (KPS) >/= 60%
* life expectancy > 9 months
* histologically proven malignant disease of the head and neck region
* lntensity Modulated RadiationTherapy (IMRT) radiotherapy
* Minimal Dose to the oral mucosa >/= 30 Gy (EQD2 w. a/ß 2)
* Simultaneous use of mouthwashes is allowed if previously prescribed by the treating physician

Exclusion Criteria:

* history of Severe oral Mucositis (SOM) due to chemotherapy within the last 3 months
* previous radiotherapy in the head-neck region
* previous cryotherapy within the last 6 weeks
* Minimal doses </=30 Gy (EQD2 w. a/ß 2)
* known history of ethylene-vinyl acetate allergy
* Simultaneous use of other forms of oral cryotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Feasability Questionnaire (regarding Patient reported tolerance of cryotherapy with Cooral ®) | up to 1 week (assessed in radiotherapy treatment period (0-10 days after baseline)
  Change in Feasability Questionnaire (regarding Patient reported tolerance of cryotherapy with Cooral ®). On this questionnaire provided to the patients at each session, they are asked to enter the break intervals and to choose a reason for the interruption from a list or to enter another reason in a provided text field. On the form there are additional question regarding the comfort of handling and wearing the device on a four scale questionnaire (the lower the score, the better the comfort of handling and wearing the device).

SECONDARY OUTCOMES:
Change in rate of OM up to 6 weeks after end of Treatment (EOT) | Assessed at baseline (0-10 days before RT) and once a week during RT and up to 6 weeks post RT.
  Change in rate of OM up to 6 weeks after end of Treatment (EOT)
Change in degree of acute OM up to 6 weeks after EOT | Assessed at baseline (0-10 days before RT) and once a week during RT and up to 6 weeks post RT.
  Change in degree of acute OM up to 6 weeks after EOT, using the CTCAE V5- scale (1 = mild to 5 = death)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Bunea, MD, Principal Investigator — University Hospital Basel, Radiotherapy and Radiation Oncology
Locations (1):
- University Hospital Basel, Radiotherapy and Radiation Oncology, Basel, Switzerland